CLINICAL TRIAL: NCT03485248
Title: Effect of Ingestion of Beet Juice on Endothelial Function, Arterial Stiffness and Muscle Oxygenation Parameters in People Living With HIV / AIDS Using Antiretroviral Therapy
Brief Title: People Living With HIV/AIDS, Nitrate, Endotelial Function, Arterial Stiffness and Skeletal Muscle Oxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Thiago Alvares, PhD, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 68923417.0.0000.5699
Record Dates: First submitted 2018-03-13; First posted 2018-04-02 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS; Arterial stiffness; Flow mediated-dilatation; Muscle oxygenation parameters; Microcirculation; Dietary Nitrate
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double- Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot juice (Active Comparator): Beetroot Juice cotaining on average 9mmol of nitrate per dose
  Interventions: Dietary Supplement: Beetroot Juice
- Placebo beet juice (Nitrate depleted) (Placebo Comparator): Beetroot juice nitrate depleted
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Beetroot Juice — 140ml of Beetroot Juice containing on avarege 9 mmol of nitrate
  Arms: Beetroot juice
Dietary Supplement: Placebo — 140ml of Beetroot Juice (nitrate free)
  Arms: Placebo beet juice (Nitrate depleted)

SUMMARY:
Administration of antiretroviral therapy has brought benefits for infective human immunodeficiency virus-1 (HIV-1)-patients, reducing the number of AIDS-related morbidity and mortality. However, it is responsible for intensifying complications triggered by the chronic inflammatory state associated with virus infection, such as cardiovascular diseases. The current study evaluated effects of single dose (140mL) of Beetroot Juice (BJ) on macro and microvascular endothelial function in HIV-1-patients undergoing antiretroviral terapy, once BJ was shown to be effective in improving these physiological parameters in uninfected individuals.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection for a period of 1 year or greater
* Regular use of high-potency antiretroviral therapy for at least one year

Exclusion Criteria:

* Individuals who are physically active
* Individuals who are allergic to some component of beet
* Individuals who use nutritional and / or pharmacological ergogenics
* Individuals receiving antibiotics or who have osteomioarticular problems

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Skeletal Muscle Oxygenation | Baseline and approximately after 150 minutes of beetroot juice consumption
  Changes in skeletal muscle oxygenation in response to exercise will be evaluated by using a near-infrared spectroscopy device.
Brachial artery flow-mediated dilatation | Baseline and approximately after 150 minutes of beetroot juice consumption
  The brachial artery flow-mediated dilation will be evaluated by using an ultrasound device.

SECONDARY OUTCOMES:
Urinary nitrate concentrations | Baseline and approximately 30, 90, and 150 minutes after beetroot juice consumption
  Analysis of nitrate in urine will be performed by using high-performance liquid chromatography system.

CONTACTS AND LOCATIONS:
Locations (1):
- DST / AIDS and Viral Hepatitis Program of Macaé, Macaé, Rio de Janeiro, Brazil